CLINICAL TRIAL: NCT00912171
Title: Efficacy of Oral Leukotriene in Long Term Therapy of Mild and Moderate Obstructive Sleep Apnea Syndrome (OSAS) in Children
Brief Title: Efficacy of Oral Leukotriene in Long Term Therapy of Mild and Moderate Obstructive Sleep Apnea Syndrome in Children
Acronym: SB-OSAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Filippo Bernardi, Associate Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 118/2007/O/Sper
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: obstructive sleep apnea syndrome; snoring; adenotonsillar hypertrophy; polysomnography; intranasal steroids; Anti-leukotrienes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring | interventions — Budesonide; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nasal steroid (Active Comparator)
  Interventions: Drug: budesonide (Aircort 50 nasal spray)
- Anti-leukotrienes (Active Comparator)
  Interventions: Drug: montelukast (Singulair)
- Nasal steroid + anti-leukotrienes (Active Comparator)
  Interventions: Drug: budesonide (Aircort 50 nasal spray); Drug: montelukast (Singulair)

INTERVENTIONS:
Drug: budesonide (Aircort 50 nasal spray) — 50 mcg per nostril once daily for cycles of 21 days with a break of 7 days for 6 months
  Other Names: Aircort 50 nasal spray
  Arms: Nasal steroid; Nasal steroid + anti-leukotrienes
Drug: montelukast (Singulair) — Daily administration in 4 mg chewable tablet for children younger than 6 years or in 5 mg tablet for children 6 years and older
  Other Names: Singulair
  Arms: Anti-leukotrienes; Nasal steroid + anti-leukotrienes

SUMMARY:
The aim of the project is to evaluate whether therapy with leukotriene may be a valid therapeutic approach in children with adenotonsillar hypertrophy and with mild and moderate obstructive sleep apnea syndrome (OSAS) and to evaluate whether leukotriene is less, equally or more efficient than nasal steroid.

DETAILED DESCRIPTION:
The aim of the project is to evaluate whether leukotriene is less, equally or more efficient than nasal steroid in children with adenotonsillar hypertrophy and with mild and moderate OSAS checking if leukotriene administrated for 24 weeks improves overnight oximetry, polysomnography and checking if leukotriene as anti-inflammatory of upper airway really reduces the tonsils and adenoids dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild (RDI 3- <5) or moderate obstructive apneas (RDI 5-8) by overnight polysomnographic evaluation with 4 channels EEG
* Adenotonsillar hypertrophy Friedman score's II-III-IV°

Exclusion Criteria:

* Neuromuscular, gastrointestinal, neurological diseases and syndromes of malformations
* Use of leukotrienes and/or nasal and oral steroids in the 4 weeks preceding the initial sleep study
* Acute upper respiratory tract infections
* Adenotonsillectomy

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Nocturnal polysomnography in the first visit compared with Nocturnal polysomnography in the last visit in patient with Montelukast treatment: | 1 year

SECONDARY OUTCOMES:
To evaluate the clinical upper airway patency during the night in the patients with history of allergic rhinitis compared with the patients without history of allergic rhinitis first and after the treatment for OSAS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Bernardi, Professor, Principal Investigator — University of Bologna
Locations (1):
- Department if Pediatrics, Hospital S. Orsola-Malpighi , University of Bologna, Bologna, Italy

REFERENCES:
- [Background] Gozal D, Crabtree VM, Sans Capdevila O, Witcher LA, Kheirandish-Gozal L. C-reactive protein, obstructive sleep apnea, and cognitive dysfunction in school-aged children. Am J Respir Crit Care Med. 2007 Jul 15;176(2):188-93. doi: 10.1164/rccm.200610-1519OC. Epub 2007 Mar 30. PMID 17400731
- [Background] Goldbart AD, Krishna J, Li RC, Serpero LD, Gozal D. Inflammatory mediators in exhaled breath condensate of children with obstructive sleep apnea syndrome. Chest. 2006 Jul;130(1):143-8. doi: 10.1378/chest.130.1.143. PMID 16840394
- [Background] Gozal D, Kheirandish-Gozal L. Sleep apnea in children--treatment considerations. Paediatr Respir Rev. 2006;7 Suppl 1:S58-61. doi: 10.1016/j.prrv.2006.04.174. Epub 2006 Jun 5. PMID 16798597
- [Background] Kheirandish L, Goldbart AD, Gozal D. Intranasal steroids and oral leukotriene modifier therapy in residual sleep-disordered breathing after tonsillectomy and adenoidectomy in children. Pediatrics. 2006 Jan;117(1):e61-6. doi: 10.1542/peds.2005-0795. PMID 16396849
- [Background] Goldbart AD, Goldman JL, Veling MC, Gozal D. Leukotriene modifier therapy for mild sleep-disordered breathing in children. Am J Respir Crit Care Med. 2005 Aug 1;172(3):364-70. doi: 10.1164/rccm.200408-1064OC. Epub 2005 May 5. PMID 15879419